CLINICAL TRIAL: NCT00577694
Title: A Nonrandomized Dose-escalation Study of Clofarabine in Combination With Gemtuzumab Ozogamicin for Relapsed/Refractory Acute Myeloid Leukemia (AML) for Patients Less Than 60 Years-old
Brief Title: Clofarabine and Gemtuzumab in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: funding unavailable
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0708; P30CA016086 (NIH); CDR0000580801 (Other: PDQ number); UNC-LCCC-07-1222
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Clofarabine; Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm study (Other): 1
  Interventions: Drug: clofarabine; Drug: gemtuzumab ozogamicin

INTERVENTIONS:
Drug: clofarabine — Intravenous, 20mg/m2, Days 1, 2, 3, 4 and 5; 2 cycles
  Other Names: Clolar
Drug: gemtuzumab ozogamicin — Intravenous, 3mg/m2, Day 1, one cycle
  Other Names: Mylotarg

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as clofarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as gemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving clofarabine together with gemtuzumab may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of clofarabine when given together with gemtuzumab in treating patients with relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify the maximum tolerated dose and dose-limiting toxicities of clofarabine when administered with gemtuzumab ozogamicin in patients with refractory acute myeloid leukemia (AML) or with AML that has relapsed within 1 year after cytarabine-containing therapy.

Secondary

* Estimate the rates of complete response and/or partial complete response with incomplete platelet recovery in patients treated with this regimen.
* Estimate the duration of remission in patients treated with this regimen and not proceeding to high-dose therapy and allogeneic stem cell transplantation.
* Estimate the frequency with which patients enrolled on this study proceed to allogeneic or autologous blood or bone marrow stem cell transplantation.

OUTLINE: This is a dose-escalation study of clofarabine.

Patients receive induction therapy comprising clofarabine IV on days 1-5 and gemtuzumab ozogamicin IV over 2 hours on days 1, 4, and 7 during course 1 only. Beginning in course 2, after blood counts recover, patients receive consolidation therapy comprising clofarabine IV on days 1-5. Consolidation treatment repeats upon blood count recovery for up to 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients in remission after consolidation therapy are followed monthly for the first 6 months, and then every 3-4 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML) meeting 1 of the following criteria:

  * Refractory disease, defined as persistent or progressive disease after ≥ 2 induction regimens, including ≥ 1 course of high-dose cytarabine (ARA-C)
  * Relapsed disease that has recurred within 1 year of an ARA-C-containing chemotherapy regimen
* No CNS disease requiring radiotherapy

  * Patients with neurological symptoms must undergo a lumbar puncture and a CT scan or MRI of the brain to exclude brain metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Total bilirubin ≤ 2.0 times upper limit of normal (ULN)
* ALT and AST ≤ 2.0 times the ULN
* Serum creatinine ≤ 1.0 mg/dL OR glomerular filtration rate > 60 mL/min
* INR ≤ 1.5 and aPTT within ULN

  * Patients receiving anticoagulation therapy (e.g., warfarin or heparin) are eligible provided anticoagulation therapy can be discontinued or changed to parenteral medications while the platelet count is less than 50,000/mm³
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent active second primary malignancy (excluding superficial, non-invasive skin cancers)
* No active bleeding diathesis, not including closely monitored therapeutic anticoagulation
* No cardiac disease, including any of the following:

  * New York Heart Association class II-IV congestive heart failure
  * Unstable angina (i.e., anginal symptoms at rest)
  * New onset angina (i.e., began within the past 3 months)
  * Myocardial infarction within the past 6 months
* No active clinically serious infection > grade 2
* No cerebrovascular accident, including transient ischemic attacks, within the past 6 months
* No pulmonary hemorrhage ≥ grade 2 within the past 4 weeks
* No other hemorrhage or bleeding event ≥ grade 3 within the past 4 weeks
* No known HIV infection or chronic hepatitis B or C
* No serious non-healing wound or ulcer
* More than 4 weeks since prior significant traumatic injury
* No prior history of sinusoidal obstructive syndrome (veno-occlusive disease)

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior major surgery or open biopsy
* More than 100 days since any prior hematopoietic stem cell transplant
* No concurrent treatment with any other investigational agent for AML

  * Intrathecal chemotherapy administration is allow for central nervous system leukemic infiltration
* No prior allogeneic stem cell transplant within the past 100 days, with active graft-versus-host disease (GVHD) of any grade, or exposure to immynosuppression for GVHD or prophylaxis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2007-11; Primary Completion 2010-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of clofarabine | 3 years

SECONDARY OUTCOMES:
Rate of complete response and/or partial complete response with incomplete platelet recovery | 3 years
Duration of remission | 5 years
Frequency of patients proceeding to allogeneic or autologous blood or bone marrow stem cell transplantation | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Shea, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States